CLINICAL TRIAL: NCT03771495
Title: What Are the Immediate Effects of Passive Hip Joint Mobilization on Hip Abductor/External Rotator Muscle Strength in Patients With Anterior Knee Pain and Impaired Hip Function
Brief Title: The Immediate Effects of Passive Hip Joint Mobilization on Hip Muscle Strength in Patients With Anterior Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: G Pflügler 09-18
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Anterior Knee Pain Syndrome; Patellofemoral Pain Syndrome
Keywords: mobilization; muscle strength; hip abductors; hip external rotators
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Joint Mobilization (Experimental): passive accessory movement on femur in anterior/posterior direction, grade III for four minutes and passive physiological movement of the most restricted hip joint movement, grade III for one minute (without pain), and a verbal education of hypothesized underlying effect mechanisms.
  Interventions: Other: Joint Mobilization
- Laying on of Hands (Sham Comparator): grade I, very small amplitude without encountering any tissue resistance for five minutes, thus effectively a Laying on of Hands, with a verbal education of hypothesized underlying effect mechanisms.
  Interventions: Other: Laying on of Hands

INTERVENTIONS:
Other: Joint Mobilization — Manual Therapy Intervention, commonly used by physiotherapists
  Arms: Hip Joint Mobilization
Other: Laying on of Hands — Sham Hip Joint Mobilization
  Arms: Laying on of Hands

SUMMARY:
The aim of the study is to assess the immediate effects of passive hip joint mobilisation (in comparison to a sham mobilisation) on eccentric hip abductor/external rotator muscle strength on the basis of manual muscle testing with a hand-held-dynamometer within a double-blinded cross-over study design. Patients with anterior knee pain and signs of impaired hip function will be recruited in Vienna and surrounding area, measurements/data collection will be conducted by two experienced physiotherapists in a physiotherapy group practice in 1150 Vienna.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis: anterior knee pain
* Prescription for physiotherapeutic treatment of anterior knee pain
* signs of functional hip impairment:
* impaired hip kinematics during single leg squat
* reduced passive hip joint mobility in comparison to the other, unaffected side
* manually weak tested hip abductors/external rota-tors in comparison to the other, unaffected side

Exclusion Criteria:

* intraarticular knee pathology
* preceding trauma/operation of lower extremity on affected side
* spinal disorders associated with low back pain, lumbar referred pain or nerve root irritation
* severe and/or recurring ankle sprains in recent history (significant enough, that it required a period of immobilization)
* other relevant comorbidities such as neurologic/rheumatologic/psychiatric diseases, osteoporosis and malign disorders
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | 10 minutes
  muscle strength data obtained from torque measurements of the hip abductor/external rotator muscles of participants before and after intervention via manual muscle testing (using a hand-held dynamometer)

CONTACTS AND LOCATIONS:
Overall Officials: Sionnadh McLean, Study Director — Sheffield Hallam University
Locations (1):
- Praxisgemeinschaft "Bewegungsoase", Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pfluegler G, Borkovec M, Kasper J, McLean S. The immediate effects of passive hip joint mobilization on hip abductor/external rotator muscle strength in patients with anterior knee pain and impaired hip function. A randomized, placebo-controlled crossover trial. J Man Manip Ther. 2021 Feb;29(1):14-22. doi: 10.1080/10669817.2020.1765625. Epub 2020 May 26. PMID 32452284

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT03771495/Prot_SAP_000.pdf